CLINICAL TRIAL: NCT05334589
Title: The Effect of Active Warming Before Total Knee Arthroplasty on Intraoperative Body Temperature and Comfort: A Randomized Control Trial
Brief Title: The Effect of Preoperative Active Warming on Intraoperative Body Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Hatice Özsoy, Lecturer, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ErsoyU
Record Dates: First submitted 2022-03-26; First posted 2022-04-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Total Knee Arthroplasty; Intraoperative Hypothermia
Keywords: Surgical nursing; Inadvertent hypothermia; Perioperative period; Active warming; Comfort

STUDY DESIGN:
Intervention Model Description: Patients were divided into intervention and control groups using the block randomization method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): Patients in the intervention group will be prewarming with a hot air blowing system for 30 minutes before the operation. The patients will continue to be warmed with a carbon fiber heating bed, which is a resistive system, during the surgery.
  Interventions: Device: Prewarming
- Control group (No Intervention): The patients will continue to be warmed with a carbon fiber heating bed, which is a resistive system, during the surgery.

INTERVENTIONS:
Device: Prewarming — When patients in the study group come to the Preoperative Care Unit (PCU), their body temperature will be measured. Patients in the study group will be placed in such a way that the 3M™ Bair Hugger™ Whole Body Blanket covers the patient's body and prewarmed with the 3M™ Bair Hugger™ Warming Unit for 30 minutes before anesthesia is given in the PCU. Heating unit temperature will be adjusted to 43°C in line with company recommendations. After the patients in the study group are warmed up for 30 minutes, the preheating process will be completed and the whole body blanket will be taken and the blankets that the clinic routinely use for each patient will be covered to cover the patients' body.
  Arms: Experimental: Intervention group

SUMMARY:
A randomized controlled study was conducted to examine the effect of active warming before total knee arthroplasty on intraoperative body temperature and comfort.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia is defined as a patient's internal temperature below 36 °C in surgical settings. All patients undergoing surgery and other invasive procedures are at risk of developing undesirable hypothermia. Both general and neuraxial anesthesia greatly impair thermoregulatory control, and as a result, unwarmed surgical patients become hypothermic. General and regional anesthesia causes undesirable hypothermia as a result of the redistribution of body temperature from the center to the periphery.

In the perioperative period, patients over 60 years of age with poor nutritional status, low core temperature before surgery, preoperative fasting and fluid deprivation before anesthesia, premedication, type of surgery, dry and cold anesthetic gases, cold intravenous fluids, flushes, blood products (cold fluids direct core temperature) Hypothermia is caused by low ambient temperature, wet skin, dressings or sheets, anesthetic agents, large open cavity or abdominal surgery, excessive blood loss, drugs used before surgery.

There are many methods to maintain the body temperature of patients (passive isolation methods) or to warm the patient (active warming methods). Passive insulation methods include heated cotton blankets, surgical drapes, and thermal suits. Active heating techniques include compressed air heaters, electric heating blankets, and heated liquids and gases.

In the literature, studies on active and passive heating methods have been found in order to prevent undesirable hypothermia. There are studies with stand-alone active heating methods (such as pressurized hot air blowing systems, heated liquids, circulating hot water systems) and combined methods. Because the results of these studies were different, a randomized controlled study was planned to investigate the effectiveness of the prewarming intervention, to support the surgical process nurses in clinical practice, and to increase the reliability of the results, before developing a procedure related to prewarming.

In the study, the effect of prewarming with a hot air blowing system before the surgical procedure on the patients who will undergo total knee arthroplasty, on the patient's body temperature during the operation and on the comfort in the early postoperative period will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered to participate in the study
* Elective surgery planned
* Patients between the ages of 18-80
* ASA I-III
* Neuroaxial anesthesia applied
* No sensory problems (hearing, vision)
* No psychiatric illness
* 18.5<BMI<39.9 kg/m2

Exclusion Criteria:

* Body temperature <36°C at the entrance to the operating room
* Preoperative body temperature <36°C
* Patients who develop complications during preheating (blood pressure rise, patients are uncomfortable with the heat, they are agitated)
* Peripheral vascular disease
* Patients with communication difficulties
* Patients with infectious disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Intraoperative body temperature | Throughout the operation (min.1 hours) (max. 2 hours)
  During the operation, the body temperature of the patients will be measured at 15-minute intervals from the beginning of the incision to the end of the operation.
  Patients' body temperature will be measured tympanically using Braun ThermoScan® 7 Age Precision®.

SECONDARY OUTCOMES:
Temperature comfort perception (before being sent to the operating room) | Before being sent to the operating room (min.15 minutes) (max.45 minutes)
  Temperature Comfort Perception Scale: Verbal Numeric Rating Scale (VNRS) between 1 and 10 (0=very comfortable; 10=very uncomfortable) will be used to objectively evaluate the temperature comfort perception of the patients.
Postoperative body temperature | Until admission to the Postanaesthesia Care Unit and sent to the clinic (min.15 minutes) (max.30 minutes)
  Body temperatures will be measured at 15-minute intervals until patients arrive at the Postanesthesia Care Unit and are sent to the clinic.
Hemodynamic parameters (Blood pressure) | From the beginning of the incision to the end of the surgery.(min.1 hours) (max. 2 hours)
  During the surgery, the blood pressure of the patients will be monitored every 15 minutes.
Hemodynamic parameters (pulse) | From the beginning of the incision to the end of the surgery.(min.1 hours) (max. 2 hours)
  During the surgery, the patients' heart rate will be monitored every 15 minutes.
Hemodynamic parameters (oxygen saturation) | From the beginning of the incision to the end of the surgery.(min.1 hours) (max. 2 hours)
  During the surgery, the oxygen saturation of the patients will be monitored every 15 minutes.
Temperature comfort perception (before sending to the clinic) | Before being sent to the clinic (min.15 minutes) (max.30 minutes)
  Temperature Comfort Perception Scale: Verbal Numeric Rating Scale (VNRS) between 1 and 10 (0=very comfortable; 10=very uncomfortable) will be used to objectively evaluate the temperature comfort perception of the patients.
Patient Comfort | Before being sent to the clinic (min.15 minutes) (max.30 minutes)
  The comfort levels of the patients who are decided to be taken from the PACU to the clinic will be measured with the Perianesthesia Comfort Scale. The highest total score that can be obtained from the scale is 144, and the lowest total score is 24. The average value is determined by dividing the total score obtained by the number of scale items, and the result is indicated in the 1-6 distribution. Low score indicates bad comfort, high score indicates good comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Özsoy, PhD Student, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Hatice Özsoy, Merkez, Burdur, Turkey (Türkiye)

REFERENCES:
- [Background] Akhtar Z, Hesler BD, Fiffick AN, Mascha EJ, Sessler DI, Kurz A, Ayad S, Saager L. A randomized trial of prewarming on patient satisfaction and thermal comfort in outpatient surgery. J Clin Anesth. 2016 Sep;33:376-85. doi: 10.1016/j.jclinane.2016.04.041. Epub 2016 Jun 3. PMID 27555196
- [Background] Rosenkilde C, Vamosi M, Lauridsen JT, Hasfeldt D. Efficacy of Prewarming With a Self-Warming Blanket for the Prevention of Unintended Perioperative Hypothermia in Patients Undergoing Hip or Knee Arthroplasty. J Perianesth Nurs. 2017 Oct;32(5):419-428. doi: 10.1016/j.jopan.2016.02.007. Epub 2016 Dec 9. PMID 28938977
- [Background] Torossian A, Van Gerven E, Geertsen K, Horn B, Van de Velde M, Raeder J. Active perioperative patient warming using a self-warming blanket (BARRIER EasyWarm) is superior to passive thermal insulation: a multinational, multicenter, randomized trial. J Clin Anesth. 2016 Nov;34:547-54. doi: 10.1016/j.jclinane.2016.06.030. Epub 2016 Jul 17. PMID 27687449